CLINICAL TRIAL: NCT05099224
Title: Effects of Mindfulness Meditation on Psychoneuroendocrinoimmunology in Nursing Students
Brief Title: Mindfulness Meditation for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Assistant Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 377/2019
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Stress Reaction; Nurse's Role
Keywords: Nursing students; Stress; C-reactive proteins; Cortisol; Mindfulness meditation
MeSH Terms: conditions — Fractures, Stress | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial (pretest-posttests, two-group, randomized design)
Who Masked: Outcomes Assessor
Masking Description: The data (questionnaire and blood samples) were collected by three research assistants with at least 10 years nursing experiences who were not involved in any other parts of the study.
  Also, the participants were randomly assigned equally to the study groups using a computerized random numbers procedure carried out by a research assistant who was not involved in any other parts of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group receiving mindfulness meditation (Experimental): The ABC standardized version of mindfulness meditation was used, which includes 5 30-minute weekly sessions of mindfulness meditation. An additional 3-hour educational workshop about the rationale and procedures of intervention was provided before the actual training sessions. The intervention was supervised by PI is an experienced practitioner who received stress-management training at the Psychology Department at Kent State University The participants were asked to sit upright in a comfortable position, place their feet on the floor, and quietly observe and reflect on internal and external stimuli such as breathing, thought, feeling, physical sensation, and sound, without reactions, judgments, or evaluations.
  Interventions: Behavioral: Mindfulness meditation
- Control group (No Intervention): Each of the control group subgroups had 10 participants. The participants were instructed to sit with their eyes closed and relax during the intervention sessions, in order to control for the nonspecific effects of trainer interaction, social interaction, attention, environment, time, and closed eyes. The timings of the control group interventions were similar to those of the experimental groups, whereby if a given experimental group intervention lasted for 30 minutes, the control group participants would be asked to sit with their eyes closed and relax for 30 minutes also.

INTERVENTIONS:
Behavioral: Mindfulness meditation — similar to the information included in arm/group descriptions
  Arms: Experimental group receiving mindfulness meditation

SUMMARY:
Mindfulness meditation was used to reduce stress and its responses such as cortisol and C-reactive protein (CRP) among healthy and ill individuals in various cultures, but their effects have not yet been studied among Jordanian nursing students, experienced tremendous stress. Thus, the purpose of study was to examine the effects of three of such intervention on perceived stress (MM) on Trait mindfulness, perceived stress, cortisol, and CRP in Jordanian nursing students. The hypothesis was " mindfulness meditation will improve trait mindfulness, perceived stress, serum cortisol and serum CRP.

Using a Randomized controlled study conducted in a large university in Jordan, 108 nursing students were randomly assigned to experimental and control groups equally. The experimental group participated in 5 30-minute weekly sessions of mindfulness meditation. Trait mindfulness, perceived stress, serum cortisol, and CRP were measured at baseline and end of intervention.

DETAILED DESCRIPTION:
Introduction Like nursing students in other countries, nursing students in Jordan have reported high stress, influencing students' health, academic performance, attrition, and ability to care for patients and themselves. Previous studies have shown that stress can negatively impact the body. Specifically, the immune system can be negatively impacted by the activation of the hypothalamic-pituitary-adrenal (HPA) system (e.g. cortisol). Elevated cortisol increases the release of pro-inflammatory factors such as C-reactive protein (CRP), found to be associated with a variety of chronic illnesses. Mindfulness meditation is a mind-body therapy that has been gaining increasing attention in the recent literature and has demonstrated promising results across different populations and settings. In Jordan, there is a lack of evidence related to the effectiveness of mindfulness meditation on stress and its physiological indices such as cortisol and CRP in Jordanian people generally and nursing students specifically. Thus, the aim was to examine the effects of three of such intervention on perceived stress (MM) on Trait mindfulness, perceived stress, cortisol, and CRP in Jordanian nursing students.

Participants and Setting The study sample included undergraduate nursing students who were selected using convenience sampling from Jordan University of Science and Technology (JUST).

Sample Size Calculation G* Power software 3.1 was used to calculate the required sample size, given a MANOVA test, an alpha of .05, power of 0.95, number of dependent variables of 4, number of groups of 2, and effect size of 0.25. A sample size of 80 was calculated, and an attrition rate of 35% was added based on a previous study with variables similar to those of the present study. Therefore, this resulted in a final total sample size of 108 participants.

Procedure First, approval from the institutional review board at JUST was obtained. After obtaining permission from the dean of the nursing college at JUST and the students' instructors, the PI visited the students in their classrooms. After the students' lecture had finished, the PI made an announcement explaining the study title and objectives and asked any students who were interested in participating to contact him either on the phone number assigned for the purposes of the study or via email. The PI arranged an initial meeting to meet with students who were interested in participating, which was to be held on another day in a private room at the university. At this meeting, the PI informed the students of the study objectives, risks, and benefits, in addition to answering the students' questions and assuring them that all collected data would be kept confidential. The students were also assured that they had the full right to refuse or discontinue participation at any time and that such refusal or discontinuation would not affect their academic achievement in any way. At the same meeting, informed consent was obtained from participants who agreed to participate and who met the eligibility criteria. After that, the participants were randomly assigned equally to the study groups using a computerized random numbers procedure carried out by a research assistant who was not involved in any other parts of the study. Finally, the dates and times of the sessions were determined.

In the 2-hour educational session, baseline measurements of the study variables were taken. Then, the PI delivered a PowerPoint presentation for the participants in each subgroup, as previously explained. At the end of the workshop, to avoid experimental contamination, the participants in each experimental group were asked not to share any information related to the intervention with the participants in the control group.

The actual training sessions were introduced to the participants in the experimental groups by the PI based on the ABC relaxation theory's guidelines and protocols. Based on the ABC Relaxation Theory, at least two, and preferably five, weekly sessions of actual mind-body training should be provided to evoke relaxation and optimize health. The sessions were held in a private, quiet, comfortable, and spacious room at the university. As previously mentioned, the dependent variables were measured twice, at baseline and at the end of the intervention (i.e., In the next morning after the 5th session).

Various strategies were followed to decrease measurement errors that could potentially be affected by variations in the data collection procedure. For example, filling out the questionnaire may be stressful for some subjects, hence influencing the objective measures. Therefore, the self-report measures were completed after the physical measures were taken. Also, all of the study measures in the intervention and control groups were taken in similar conditions, including similar room temperature and environment. In addition, quiet environments were maintained, with a "Do Not Disturb" sign placed on the doors of the rooms during the interventions and data collection.

Statistical Analysis Statistical analysis was conducted using SPSS software (version 25). Descriptive statistics were used to describe the sample. The sample and study variables were described by measures of central tendency and dispersion appropriate to the level of measurement. Initial independent t-tests and Chi-squared tests were conducted to ensure that the randomization across the covariates was successful, and one-way MANOVA was used to test the study hypotheses. Post hoc one-way ANOVAs were run to examine if there were significant differences in each of the dependent variables between the study groups. Due to multiple testing, the p-value was adjusted by dividing the p value of .05 by 4 (i.e., the number of dependent variables), with a level of .0125 considered as the level of significance for the ANOVA tests.

ELIGIBILITY:
Inclusion Criteria:

* The study sample included undergraduate nursing students who were aged 18 years or over and taking a clinical course

Exclusion Criteria:

* Students were excluded if they were practicing any type of relaxation techniques or taking hypnotics, sedatives, anxiolytics, anti-depressants, or anti-hypertensive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Trait Mindfulness | 6 weeks
  Trait mindfulness was measured using the Arabic version of the Mindful Attention Awareness Scale (MAAS) (28), which is a one-dimensional scale that includes 15 items measured on a six-point Likert-type scale ranging from 1 (almost always) to 6 (almost never). The total possible score ranges between 15 and 90, with higher scores indicating higher levels of trait mindfulness. The original scale has been shown to have strong psychometric properties when validated among college students (28). Further, the Arabic version of this scale has been shown to have excellent internal consistency and convergent validity for use among Arab populations (29). In the current study, the Cronbach's alpha for the Arabic version of the MAAS was .79, indicating good internal consistency.
Perceived stress | 6 weeks
  The Perceived Stress Scale (PSS) (30) is used to measure the degree to which situations in one's life are appraised as stressful (unpredictable, uncontrollable, and overloaded). The scale comprises 10 items which are measured on a 5-point Likert scale (0=never, 4= very often) and which are relatively free of content specific to any subpopulation group. The total possible score ranges from 0 to 40, with higher scores indicating higher levels of perceived stress (30). The PSS has been validated for use among college students, with internal consistency coefficients ranging from .84 to 36 and a test-retest reliability of .85 (30). The Arabic version of the PSS, which was used in the present study, has been shown to have adequate reliability and validity and is considered a suitable instrument for assessing perceived stress among Arab populations (31). In the current study, the Cronbach's alpha for the Arabic version of the PSS was .81, indicating good internal consistency.
Serum cortisol | 6 weeks
  The ELISA method has been found to be accurate, sensitive, specific, and precise in terms of determining the plasma concentration of cortisol (32). In the current study, the ELISA kit and protocols were used to analyze the blood sample for the serum cortisol (CEA462Ge) . Three research assistants with at least 10 years of experience collected 10 mL blood samples via venipuncture both at baseline and next day morning after the last session, between 8:30-9:30 AM. The results were read using a SYNERGY (HTZ) multi-mode reader, connected to a computer which showed each reading value. The participants were asked to avoid caffeine consumption on the days of data collection. To decrease venipuncture-related pain during blood sampling, the EMLA cream was used, as it has been found effective in decreasing venipuncture-related pain among different populations (33).
Serum CRP | 6 weeks
  The ELISA kit and protocols were used to analyze the blood sample for the serum CRP (Cat no: SEA821Hu) . Three research assistants with at least 10 years of experience collected 10 mL blood samples via venipuncture both at baseline and next day morning after the last session, between 8:30-9:30 AM. The results were read using a SYNERGY (HTZ) multi-mode reader, connected to a computer which showed each reading value. The participants were asked to avoid caffeine consumption on the days of data collection. To decrease venipuncture-related pain during blood sampling, the EMLA cream was used, as it has been found effective in decreasing venipuncture-related pain among different populations (33).

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Hossam AlHawatmeh, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster K, Roche M, Giandinoto JA, Platania-Phung C, Furness T. Mental health matters: A cross-sectional study of mental health nurses' health-related quality of life and work-related stressors. Int J Ment Health Nurs. 2021 Jun;30(3):624-634. doi: 10.1111/inm.12823. Epub 2020 Dec 5. PMID 33280229
- [Background] Al-Zayyat AS, Al-Gamal E. Perceived stress and coping strategies among Jordanian nursing students during clinical practice in psychiatric/mental health courses. Int J Ment Health Nurs. 2014 Aug;23(4):326-35. doi: 10.1111/inm.12054. Epub 2013 Dec 25. PMID 24372812
- [Background] Labrague LJ, McEnroe-Petitte DM, De Los Santos JAA, Edet OB. Examining stress perceptions and coping strategies among Saudi nursing students: A systematic review. Nurse Educ Today. 2018 Jun;65:192-200. doi: 10.1016/j.nedt.2018.03.012. Epub 2018 Mar 21. PMID 29602137
- [Background] Chaabane S, Chaabna K, Bhagat S, Abraham A, Doraiswamy S, Mamtani R, Cheema S. Perceived stress, stressors, and coping strategies among nursing students in the Middle East and North Africa: an overview of systematic reviews. Syst Rev. 2021 May 5;10(1):136. doi: 10.1186/s13643-021-01691-9. PMID 33952346
- [Background] Kinlein SA, Karatsoreos IN. The hypothalamic-pituitary-adrenal axis as a substrate for stress resilience: Interactions with the circadian clock. Front Neuroendocrinol. 2020 Jan;56:100819. doi: 10.1016/j.yfrne.2019.100819. Epub 2019 Dec 19. PMID 31863788
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] Sousa GM, Lima-Araujo GL, Araujo DB, Sousa MBC. Brief mindfulness-based training and mindfulness trait attenuate psychological stress in university students: a randomized controlled trial. BMC Psychol. 2021 Feb 1;9(1):21. doi: 10.1186/s40359-021-00520-x. PMID 33526085
- [Background] Bottaccioli AG, Bottaccioli F, Carosella A, Cofini V, Muzi P, Bologna M. Psychoneuroendocrinoimmunology-based meditation (PNEIMED) training reduces salivary cortisol under basal and stressful conditions in healthy university students: Results of a randomized controlled study. Explore (NY). 2020 May-Jun;16(3):189-198. doi: 10.1016/j.explore.2019.10.006. Epub 2019 Nov 14. PMID 31982328
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Rayan A, Ahmad M. The psychometric properties of the mindful attention awareness scale among Arab parents of children with autism spectrum disorder. Arch Psychiatr Nurs. 2018 Jun;32(3):444-448. doi: 10.1016/j.apnu.2018.01.001. Epub 2018 Jan 3. PMID 29784228
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Almadi T, Cathers I, Hamdan Mansour AM, Chow CM. An Arabic version of the perceived stress scale: translation and validation study. Int J Nurs Stud. 2012 Jan;49(1):84-9. doi: 10.1016/j.ijnurstu.2011.07.012. Epub 2011 Aug 17. PMID 21851941
- [Background] Levine A, Zagoory-Sharon O, Feldman R, Lewis JG, Weller A. Measuring cortisol in human psychobiological studies. Physiol Behav. 2007 Jan 30;90(1):43-53. doi: 10.1016/j.physbeh.2006.08.025. Epub 2006 Oct 19. PMID 17055006
- [Background] Fetzer SJ. Reducing venipuncture and intravenous insertion pain with eutectic mixture of local anesthetic: a meta-analysis. Nurs Res. 2002 Mar-Apr;51(2):119-24. doi: 10.1097/00006199-200203000-00008. PMID 11984382
- [Background] Smith JC. Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company; 2005 Mar 4.
- [Background] Rausch SM, Gramling SE, Auerbach SM. Effects of a single session of large-group meditation and progressive muscle relaxation training on stress reduction, reactivity, and recovery. International Journal of Stress Management. 2006 Aug;13(3):273.
- [Background] Ghoncheh S, Smith JC. Progressive muscle relaxation, yoga stretching, and ABC relaxation theory. J Clin Psychol. 2004 Jan;60(1):131-6. doi: 10.1002/jclp.10194. PMID 14692015
- [Background] Matsumoto M, Smith JC. Progressive muscle relaxation, breathing exercises, and ABC relaxation theory. J Clin Psychol. 2001 Dec;57(12):1551-7. doi: 10.1002/jclp.1117. PMID 11745596
- [Background] Knight, Erik L., et al.
- [Background] Markozannes, Georgios, et al.
- [Background] Khader YS, Alsadi AA. Smoking habits among university students in Jordan: prevalence and associated factors. East Mediterr Health J. 2008 Jul-Aug;14(4):897-904. PMID 19166173
- [Background] Khater W, Akhu-Zaheya L, Shaban I. Sources of stress and coping behaviours in clinical practice among baccalaureate nursing students. International Journal of Humanities and Social Science. 2014 Apr;4(6):194-202
- [Background] Amanvermez Y, Rahmadiana M, Karyotaki E, de Wit L, Ebert DD, Kessler RC, Cuijpers P. Stress management interventions for college students: A systematic review and metaanalysis. Clinical Psychology: Science and Practice. 2021 Aug 12
- [Background] Yanyu J, Xi Y, Huiqi T, Bangjiang F, Bin L, Yabin G, Xin M, Junhua Z, Zhitao Y, Xiaoyun C, Changsheng D. Meditation-based interventions might be helpful for coping with the Coronavirus disease 2019 (COVID-19)
- [Background] M. Virgili, Mindfulness-based interventions reduce psychological distress in working adults: a meta-analysis of intervention studies, Mindfulness 6 (2) (2015) 326-337, https://doi.org/10.1007/s12671-013-0264-0.
- [Background] de Vibe M, Solhaug I, Tyssen R, Friborg O, Rosenvinge JH, Sorlie T, Bjorndal A. Mindfulness training for stress management: a randomised controlled study of medical and psychology students. BMC Med Educ. 2013 Aug 13;13:107. doi: 10.1186/1472-6920-13-107. PMID 23941053
- [Background] Garland E, Gaylord S, Park J. The role of mindfulness in positive reappraisal. Explore (NY). 2009 Jan-Feb;5(1):37-44. doi: 10.1016/j.explore.2008.10.001. PMID 19114262
- [Background] Kabat-Zinn, Mindfulness-based interventions in context: past, present, and future, Clin. Psychol. Sci. Pract. 10 (2) (2003) 144-156, https://doi.org/10.1093/clipsy/ bpg016
- [Background] Lahtinen O, Aaltonen J, Kaakinen J, Franklin L, Hyona J. The effects of app-based mindfulness practice on the well-being of university students and staff. Curr Psychol. 2023;42(6):4412-4421. doi: 10.1007/s12144-021-01762-z. Epub 2021 May 1. PMID 33967565
- [Background] Lazarus RS, Folkman S. Stress, appraisal, and coping. Springer publishing company; 1984 Mar 15
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Chiodelli R, Mello LTN, Jesus SN, Andretta I. Effects of a brief mindfulness-based intervention on emotional regulation and levels of mindfulness in senior students. Psicol Reflex Crit. 2018 Aug 2;31(1):21. doi: 10.1186/s41155-018-0099-7. PMID 32026168
- [Background] Sanada K, Montero-Marin J, Alda Diez M, Salas-Valero M, Perez-Yus MC, Morillo H, Demarzo MM, Garcia-Toro M, Garcia-Campayo J. Effects of Mindfulness-Based Interventions on Salivary Cortisol in Healthy Adults: A Meta-Analytical Review. Front Physiol. 2016 Oct 19;7:471. doi: 10.3389/fphys.2016.00471. eCollection 2016. PMID 27807420
- [Background] Stevens BS, Royal KD, Ferris K, Taylor A, Snyder AM. Effect of a mindfulness exercise on stress in veterinary students performing surgery. Vet Surg. 2019 Apr;48(3):360-366. doi: 10.1111/vsu.13169. Epub 2019 Jan 29. PMID 30693966
- [Background] Tang YY, Tang R, Jiang C, Posner MI. Short-term meditation intervention improves self-regulation and academic performance. J Child Adolesc Behav. 2014;02
- [Background] Parsons EM, Dreyer-Oren SE, Magee JC, Clerkin EM. Evaluating the Indirect Effects of Trait Mindfulness Facets on State Tripartite Components Through State Rumination and State Experiential Avoidance. J Nerv Ment Dis. 2019 Jun;207(6):440-450. doi: 10.1097/NMD.0000000000000993. PMID 31045980
- [Background] Heckenberg RA, Eddy P, Kent S, Wright BJ. Do workplace-based mindfulness meditation programs improve physiological indices of stress? A systematic review and meta-analysis. J Psychosom Res. 2018 Nov;114:62-71. doi: 10.1016/j.jpsychores.2018.09.010. Epub 2018 Sep 22. PMID 30314581
- [Derived] Alhawatmeh HN, Rababa M, Alfaqih M, Albataineh R, Hweidi I, Abu Awwad A. The Benefits of Mindfulness Meditation on Trait Mindfulness, Perceived Stress, Cortisol, and C-Reactive Protein in Nursing Students: A Randomized Controlled Trial. Adv Med Educ Pract. 2022 Jan 13;13:47-58. doi: 10.2147/AMEP.S348062. eCollection 2022. PMID 35046747

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT05099224/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05099224/ICF_001.pdf